CLINICAL TRIAL: NCT05805176
Title: An Adjunct Study to Assess Guided ADHD Therapy for Managing the Extent and Severity of Symptoms - A Prospective, Multicenter, Open Label, Single Arm, Intervention Study to Assess Efficacy and Safety of an At-home, Game-based Digital Therapy for Treating Clinical Symptoms of Adult Patients With Attention-Deficit/Hyperactivity Disorder (ADHD)
Brief Title: An Adjunct Study to Assess Guided ADHD Therapy for Managing the Extent and Severity of Symptoms
Acronym: A-GAMES
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lumos Labs, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP-014
Record Dates: First submitted 2023-03-24; First posted 2023-04-07 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ADHD Therapy (Experimental)
  Interventions: Device: ADHD Therapy

INTERVENTIONS:
Device: ADHD Therapy — investigational game-play therapy

SUMMARY:
The objective of this study is to assess the safety and effectiveness of an at-home, game-based digital therapy for treating adult patients with Attention-Deficit/Hyperactivity Disorder (ADHD).

ELIGIBILITY:
Inclusion Criteria:

* 22-55 years of age (Cohort I) or 18-21 years of age (Cohort II)
* Confirmed ADHD diagnosis, combined or inattentive type, at Screening based on DSM-5 criteria and established via the MINI-Adult, administered by a trained clinician
* Baseline total score on the DSM 5 Inattentive Symptoms, DSM 5 Hyperactive - Impulsive Symptoms and ADHD Index subscales of the Conners' Adult ADHD Rating Scales-Investigator Rated: Long Version (CAARS-Inv:L) ≥24
* Current, stable use of an FDA approved pharmacological treatment for ADHD for at least 4 weeks prior to screening, but ADHD condition inadequately managed by that medication
* Ability to understand and speak English, follow written and verbal instructions (English), as assessed by the PI and/or Study Coordinator, and give informed consent (English)
* Have ability to connect wireless devices to a functional wireless network daily
* Have access to a computer or smart device (e.g., phone, tablet) with internet access and a Google Chrome web browser
* Ability to comply with all the testing and study requirements

Exclusion Criteria:

* Unstable/uncontrolled, comorbid psychiatric diagnosis, based on clinical interviewing, with significant current active symptoms including but not limited to posttraumatic stress disorder, schizophrenia spectrum and other psychotic disorders, bipolar disorder, autism spectrum disorder, severe obsessive-compulsive disorder, severe depressive or severe anxiety disorder, conduct disorder, or other symptomatic manifestations that in the opinion of the Investigator may confound study data/assessments
* Inadequate IQ to participate in the study as estimated by Investigator (i.e., inability to read/understand the informed consent; inability to understand how the device and therapy (games) work)
* PHQ-9 scores ≥16
* Have previously been assessed by TOVA for potential enrollment in a clinical trial.
* Have previously used a videogame-like digital therapy (e.g., Akili EndeavorRxTM) OR within the last three years, have used a cognitive or brain training platform (e.g., Peak, Brain HQ, Lumosity, Atentiv) for more than two weeks duration
* Known sensitivity to playing video games, such as headaches, dizziness, nausea
* Initiation within the last 4 weeks of behavioral therapy or neurofeedback, or planned initiation during the study. Patients who have been in behavior therapy or neurofeedback consistently for more than 4 weeks may participate provided their routine is unchanged during the course of the study. Patients planning on changing or initiating behavior therapy or neurofeedback during the course of the study will be excluded
* Patient is currently considered a suicide risk in the opinion of the Investigator, as measured by C-SSRS at screening (i.e., score of 4 or 5 on C-SSRS)
* Motor condition (e.g., physical deformity of the hands/arms; protheses) that prevents game playing as observed by the Investigator
* Recent history (within the past 12 months) of suspected alcohol or substance abuse or dependence
* Positive urine drug screen
* History of seizures (excluding febrile seizures), or significant motor or vocal tics, including but not limited to Tourette's Disorder and photo-sensitive epilepsy
* Visual acuity that cannot be corrected that prevents or negatively impacts game playing as observed by the Investigator
* Any use of psychoactive drugs (other than ADHD medication) that in the opinion of the Investigator may confound study data/assessments
* Has participated in a clinical trial within 90 days prior to screening
* Has a family member or close friend/associate also enrolled/currently participating in the same study
* Any other condition that in the opinion of the Investigator may confound study data/assessments

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 194 (Actual)
Dates: Start 2023-04-15 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Conners' Adult ADHD Rating Scales-Investigator Rated: Long Version (CAARS-Inv:L) Inattentive Symptoms subscale | Study Day 0 to Study Day 63
  The Conners' Adult ADHD Rating Scales-Investigator Rated: Long Version (CAARS-Inv:L) has 66 items with multiple subscales.

SECONDARY OUTCOMES:
Adult ADHD Self-Report Scale (ASRS) Inattentive Symptoms Subscale | Study Day 0 to Study Day 63
  The World Health Organization Adult Self-Report Scale (ASRS) symptom checklist is an 18-item tool to screen for probable ADHD in adults. The ASRS checklist asks respondents to indicate how they have felt and conducted themselves over the past 6 months in terms of frequency of inattention or hyperactivity symptoms, which are rated from 0 ("never") to 4 ("very often"). The checklist is divided into two parts and results in a "Part A" inattention subscore (range 0-36), a "Part B" hyperactivity/ impulsivity subscore (range 0-36), and a total score based on the full scale (range 0-72).
Conners' Adult ADHD Rating Scales-Investigator Rated: Long Version (CAARS-Inv:L) ADHD Symptoms Total subscale | Study Day 0 to Study Day 63
  The Conners' Adult ADHD Rating Scales-Investigator Rated: Long Version (CAARS-Inv:L) has 66 items with multiple subscales.
Sheehan Disability Scale (SDS) | Study Day 0 to Study Day 63
  The Sheehan Disability Scale is a five-item, self-rated questionnaire designed to measure the extent to which a patient's disability due to an illness or health problem interferes with work/school, social life/leisure activities, and family life/home responsibilities.

CONTACTS AND LOCATIONS:
Overall Officials: Greg Mattingly, MD, Principal Investigator — Midwest Research Group
Locations (5):
- United States (5):
  - CNS Healthcare of Jacksonville, Jacksonville, Florida
  - Accel Clinical Research Sites, Lakeland, Florida
  - Rochester Center for Behavioral Medicine (RCBM), Rochester Hills, Michigan
  - Midwest Research Group, Brentwood, Missouri
  - Hassman Research Institute, Berlin, New Jersey

IPD SHARING:
Plan to Share IPD: No